CLINICAL TRIAL: NCT03946930
Title: A Cohort Study of Cognitive Decline in Alzheimer Disease
Brief Title: Cognitive Decline in AD
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Timothy Kwok, Professor, Chinese University of Hong Kong
Other Study IDs: 2018.274
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is lack of information on the risk factors of accelerated cognitive decline in older people with Alzheimer disease (AD). The extent of neurodegeneration and white matter disease has been reported to be important factors. In addition there may be biomarkers e.g. inflammatory cytokines that can contribute to cognitive decline. The impact of care arrangement and physical activity may also be important. Insulin signaling is impaired in Alzheimer disease (AD).

We therefore propose to perform a cohort study of older people with AD. This will be based on an on-going AD registry which was designed to identify genetic biomarkers for AD. Detailed neurocognitive tests and lifestyle information are available. In addition, volumetric MRI brain scans were performed in all AD subjects. The hypothesis is that MRI brain volumes, serum biomarkers, physical activity, physical functioning are independently associated with cognitive decline in older people with AD. The objective is to identify risk factors of accelerated cognitive decline so that preventive measures can be designed to delay dependency in AD.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient Cantonese competency for cognitive test
* Clinical diagnosis of AD
* FAST test staging 3-5

Exclusion Criteria:

* Subjects who refuse blood taking procedure
* No reliable family caregiver informant (person contact at least once a month)

Ages: 65 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Subjects are recruited from the geriatric outpatient clinics or memory clinic.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-12-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-cognitive subscale ADAS-COG | 24-Months
  Cognitive assessment for dementia

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong